CLINICAL TRIAL: NCT02058966
Title: Pilot Study of the Dose Response of Entacapone on Methamphetamine Induced Interest, Mood Elevation, and Reward
Brief Title: Pilot Study of Entacapone for Methamphetamine Abuse
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Hoffman, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 8874; 1004805 (Other: OHSU InfoEd); 3986 (Other: OCTRI)
Record Dates: First submitted 2014-02-05; First posted 2014-02-11 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Methamphetamine Dependence
Keywords: Entacapone; COMT val158met; Methamphetamine
MeSH Terms: interventions — entacapone; Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo followed by Placebo (Placebo Comparator): Subjects will receive placebo, then one hour later, placebo
  Interventions: Drug: Placebo
- Placebo followed by Methamphetamine (Experimental): Subjects will receive placebo, then one hour later, methamphetamine
  Interventions: Drug: Methamphetamine; Drug: Placebo
- Entacapone followed by Placebo (Experimental): Subjects will receive entacapone, then one hour later, placebo
  Interventions: Drug: Entacapone; Drug: Placebo
- Entacapone followed by Methamphetamine (Experimental): Subjects will receive entacapone, then one hour later, methamphetamine
  Interventions: Drug: Entacapone; Drug: Methamphetamine

INTERVENTIONS:
Drug: Entacapone — Entacapone 200 mg oral dose
  Other Names: Comtam
  Arms: Entacapone followed by Methamphetamine; Entacapone followed by Placebo
Drug: Methamphetamine — Methamphetamine 20 mg oral dose
  Other Names: Desoxyn
  Arms: Entacapone followed by Methamphetamine; Placebo followed by Methamphetamine
Drug: Placebo — capsules compounded to be of similar appearance to the active drugs
  Arms: Entacapone followed by Placebo; Placebo followed by Methamphetamine; Placebo followed by Placebo

SUMMARY:
Addiction to methamphetamine is a serious health problem. There are no medications that a doctor can give someone to help them stop using methamphetamine. Entacapone (Comtan©) is a medication that could help people addicted to methamphetamine.

This study will see how entacapone works in healthy people who are given methamphetamine. We think that the study drug will be well tolerated, and that it will prevent some of the effects of methamphetamine that make it so addictive. We also want to see how differences in people's genes may cause differences in the ways the study drug and methamphetamine work for them.

The study has six total visits. The first visit is for screening. Tests and procedures will make sure it is safe for subjects to participate.

The second visit is a familiarization day. Subjects will receive methamphetamine, but no entacapone. This is done to make sure they can tolerate the drug and recognize its effects before being given a second drug on the same day. Subjects will take surveys and computer tests to see how the medications change mood, thinking, and liking the drug.

The final four visits are the actual study days. Subjects will be randomly assigned (like the flip of a coin) to the different ways to get either 1) study medication or placebo (placebo contains no active study medication) and then 2) methamphetamine or placebo. Subjects will be in all four groups during the study, which means that each day a subject will get a different group.

ELIGIBILITY:
Inclusion Criteria:

* No history of pre-existing physical (including cardiovascular) illness
* No history of drug abuse or dependence
* Ability to read and write English
* Have had at least one exposure to a stimulant (e.g. cocaine, methamphetamine, ecstasy, methylphenidate or any medication in the stimulant class) in their lifetime

Exclusion Criteria:

* Pregnant
* Taking any psychotropic medication
* Meeting DSM-IV criteria for active substance abuse or dependence
* On any stimulant medication
* History or current hypertension (BP > 140/90 mm Hg) or systolic hypotension (SBP < 90 mm Hg)
* Subjects with resting pulse rate > 90/min
* Any active medical illness
* Family history of abnormal heart rhythms, or sudden cardiac death
* Subjects who anticipate they may require the emergent use of epinephrine (such as an Epi-Pen®) for the treatment of severe allergic reactions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Fellers, MD, Principal Investigator — Oregon Health and Science University; William F Hoffman, MD, PhD, Principal Investigator — VA Portland Healthcare System
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study staff screened 80 subjects over the phone between June 2014 to June 2016 at a clinical hospital in Portland, OR.
Pre-assignment Details: 51 subjects failed the pre-screen primarily due to history of substance use disorder, time commitment conflicts, or unwilling to take methamphetamine. 14 of 29 subjects completed first randomization. Of the 29, 6 declined to participate, 4 did not meet inclusion criteria, 1 was excluded due to an adverse event, and 6 dropped out.
Groups:
- All Subjects: Subjects will get either entacapone or placebo, then one hour later, either methamphetamine or placebo.
  Placebo: capsules compounded to be of similar appearance to the active drugs
  Entacapone: Entacapone 200 mg oral dose
  Methamphetamine: Methamphetamine 20 mg oral dose
  The research pharmacy will assign randomization; they have no contact with the subjects or clinical staff involved in direct subject care so this medication combination could occur at any of the 4 randomization visits.
Period: Open-Label Methamphetamine
Arm/Group | All Subjects
Started | 19
Received Methamphetamine | 18
Completed | 18
Not Completed | 1
Not completed — Adverse Event | 1
Period: First Intervention
Arm/Group | All Subjects
Started (3 subjects dropped out between Open-Label Methamphetamine and First Intervention.) | 15
Received Placebo-Placebo | 3
Received Placebo-Meth | 4
Received Entacapone-Placebo | 2
Received Entacapone-Meth | 5
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Intervention
Arm/Group | All Subjects
Started (1 subject dropped out between First and Second Intervention.) | 13
Received Placebo-Placebo | 2
Received Placebo-Meth | 2
Received Entacapone-Placebo | 6
Received Entacapone-Meth | 3
Completed | 13
Not Completed | 0
Period: Third Intervention
Arm/Group | All Subjects
Started (1 subjects dropped out between Second and Third Intervention.) | 12
Received Placebo-Placebo | 4
Received Placebo-Meth | 4
Received Entacapone-Placebo | 1
Received Entacapone-Meth | 3
Completed | 12
Not Completed | 0
Period: Fourth Intervention
Arm/Group | All Subjects
Started | 12
Received Placebo-Placebo | 4
Received Placebo-Meth | 3
Received Entacapone-Placebo | 3
Received Entacapone-Meth | 2
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline measurements were taken during each randomization visit before participant received any drug treatment. Baseline measurements were then averaged over the 4 randomization visits.
Groups:
- All Participants: Participants who completed all four study arms including:
  1. Placebo followed by Placebo
  2. Placebo followed by Methamphetamine (20 mg)
  3. Entacapone (200 mg) followed by Placebo
  4. Entacapone (200 mg) followed by Methamphetamine (20 mg)
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Effect of Entacapone on Methamphetamine-induced Mood
Description: Profile of Mood States is a 65 item questionnaire using a Likert rating scale to assess transient, distinct moods. The questionnaire contains 65 words/statements that describe feelings people have. The test requires you to indicate for each word or statement how you have been feeling in the past week including today. A Total Mood Disturbance score is calculated by adding scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the Vigour score. The Total Mood Disturbance scale ranges from -32 to 200 with lower scores indicative of people with more stable mood profiles.
Time Frame: Measurements acquired before drug ingestion (baseline) then hourly for 4 hours. The peak interaction effect of entacapone and methamphetamine occurs 1 hour after ingestion, therefore the reported values are from this timepoint.
Population: The analysis population includes only the 12 subjects that completed each intervention of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Baseline measurements were taking for each subject before drug intervention during each of the 4 visits then averaged over the 4 visits. Baseline measurements reported here are averaged across all subjects.
Arm/Group | Baseline | Placebo Followed by Placebo | Placebo Followed by Methamphetamine | Entacapone Followed by Placebo | Entacapone Followed by Methamphetamine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
units on a scale | 12.500 (8.187) | 13.750 (9.037) | 7.500 (4.166) | 9.833 (4.783) | 8.750 (4.309)

2. Primary Outcome: Effect of Entacapone on Subjective Effects of Methamphetamine
Description: The subjective effects of the study drug were evaluated with the Addiction Research Center Inventory (ARCI-49), a 49 item questionnaire consisting of true/false items. True items receive a score of 1 if answer is 'True', false items receive a score of 1 if answer is 'False'. No points are given when answer is opposite to scoring direction. There are 5 subscales: Morphine Benzedrine group scale to measure euphoria (range: 0-16 with higher numbers indicating more euphoria), A Lysergic Acid Diethylamide group scale to estimate dysphoria and agitation (range: 0-14 with higher scores indicating more dysphoria), a Pentobarbital Chlorpromazine Alcohol group scale to measure sedation (range: 0-15 with higher scores indicating more sedation), and a Benzedrine group scale and an Amphetamine Scale to assess stimulant effects (range: 0-13 and 0-11, respectively, with higher scores indicating higher stimulant effects) .
Time Frame: as for outcome 1
Population: The analysis population includes only the 12 subjects that completed each arm, or intervention, of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Placebo Followed by Placebo | Placebo Followed by Methamphetamine | Entacapone Followed by Placebo | Entacapone Followed by Methamphetamine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
units on a scale
  Morphine Benzedrine | 1.9375 (2.6610) | 1.8333 (2.8868) | 7.9167 (5.9308) | 2.5833 (4.1000) | 6.9167 (6.2879)
  Lysergic Acid Diethylamide | 3.0625 (1.1923) | 3.25 (1.1382) | 4.75 (2.0944) | 3.25 (1.1382) | 3.8333 (1.3371)
  Pentobarbital Chlorpromazine Alcohol | 4.8125 (2.5066) | 5.0000 (2.9233) | 1.5833 (1.8320) | 4.0833 (2.8110) | 2.0000 (2.1320)
  Benzedrine | 4.9583 (1.4869) | 5.1667 (2.0817) | 8.6667 (3.6013) | 5.3333 (2.1462) | 7.8333 (3.7376)
  Amphetamine | 2.0000 (1.8451) | 2.1667 (2.4802) | 5.9167 (3.4499) | 2.5833 (2.6097) | 5.5833 (4.0104)

3. Primary Outcome: Effect of Entacapone on Methamphetamine-induced Stimulation
Description: The Global Rating of Stimulation is a 1-item question "I feel light-headed, restless, or speeded-up" in which the participant is asked to circle one answer on a scale from 0-4, 0 is 'normal', 1 is 'slightly', 2 is 'moderately', 3 is 'very much', and 4 is 'extremely'. Whichever number they circled is their reported score. A higher score is indicative of a greater stimulating effect.
Time Frame: as for outcome 1
Population: The analysis population includes only the 12 subjects that completed each arm, or intervention, of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Placebo Followed by Placebo | Placebo Followed by Methamphetamine | Entacapone Followed by Placebo | Entacapone Followed by Methamphetamine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
units on a scale | 0.1667 (0.5586) | 0.1667 (0.5774) | 1.4167 (1.1645) | 0.4167 (0.9003) | 1.3333 (1.1547)

4. Secondary Outcome: Cognitive Function
Description: Two computer tests were administered to measure how each medication intervention effects cognitive functioning. The tests administered included the Rapid Visual Information Processing Task (RVIPT), a 6 minute test of sustained attention in which participants are requested to detect target sequences of digits and the Digit Symbol Substitution Task (DSST), a 2 minute test of psychomotor speed and sustained attention consisting of digit-symbol pairs followed by a list of digits where the subject identifies the symbol that corresponds to each digit as fast as possible. The number of correct responses within the allowed time is measured. Higher scores on both tasks indicate better performance.
Time Frame: as for outcome 1
Population: The analysis population includes only the 12 subjects that completed each arm, or intervention, of the study.
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Baseline | Placebo Followed by Placebo | Placebo Followed by Methamphetamine | Entacapone Followed by Placebo | Entacapone Followed by Methamphetamine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
number of correct answers
  Rapid Visual Information Processing Task | 38.813 (11.230) | 40.500 (13.215) | 41.333 (11.073) | 42.583 (10.423) | 40.083 (10.396)
  Digital Symbol Substitution Task | 73.167 (17.765) | 72.000 (20.662) | 71.167 (27.788) | 72.750 (14.973) | 72.750 (15.004)

ADVERSE EVENTS:
Groups:
- Open-label Methamphetamine: Subject will receive one dose of open-label methamphetamine 20 mg oral dose on their second visit, the familiarization visit.
- Placebo-Placebo: Subjects will receive placebo, then one hour later, placebo
  Placebo: capsules compounded to be of similar appearance to the active drugs
- Placebo-Meth: Subjects will receive placebo, then one hour later, methamphetamine
  Placebo: capsules compounded to be of similar appearance to the active drugs
  Methamphetamine: Methamphetamine 20 mg oral dose
- Entacapone-Placebo: Subjects will receive entacapone, then one hour later, placebo
  Placebo: capsules compounded to be of similar appearance to the active drugs
  Entacapone: Entacapone 200 mg oral dose
- Entacapone-Meth: Subjects will receive entacapone, then one hour later, methamphetamine
  Methamphetamine: Methamphetamine 20 mg oral dose
  Entacapone: Entacapone 200 mg oral dose
Arm/Group | Open-label Methamphetamine | Placebo-Placebo | Placebo-Meth | Entacapone-Placebo | Entacapone-Meth
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/13 | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/13 | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 1/19 | 0/13 | 0/13 | 0/12 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Methamphetamine (N=19) | Placebo-Placebo (N=13) | Placebo-Meth (N=13) | Entacapone-Placebo (N=12) | Entacapone-Meth (N=13)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One subject's blood pressure reached 180/100 after ingesting Methamphetamine 20 mg pill but was in the 160s/90s for two hours before normalizing. This subject was removed from the study after this incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No